CLINICAL TRIAL: NCT01723514
Title: Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 334 in Healthy Subjects and in Migraine Patients
Brief Title: Ascending Multiple-Doses of Erenumab (AMG 334) in Healthy Adults and in Migraine Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20101268; 2012-003594-26 (EudraCT Number)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erenumab (Experimental): Healthy participants and participants with migraine received subcutaneous doses of erenumab on days 1, 29 and 57.
  Interventions: Drug: Erenumab
- Placebo (Placebo Comparator): Healthy participants and participants with migraine received subcutaneous doses of placebo on days 1, 29 and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erenumab — Administered by subcutaneous injection once a month
  Other Names: AMG-334; Aimovig™
  Arms: Erenumab
Drug: Placebo — Administered by subcutaneous injection once a month
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether erenumab is safe and well tolerated in healthy adults and migraine patients. As part of the secondary objectives, this study will be conducted to characterize the pharmacokinetic (PK) profile of erenumab after multiple subcutaneous (SC) doses in healthy adults and migraine patients, as well as to characterize the effect of erenumab on the capsaicin induced increase in dermal blood flow after multiple SC doses in healthy adults and migraine patients.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female subjects, as well as male or female subjects with migraines between 18 and 55 years of age, inclusive, with no history or evidence of clinically relevant medical disorders as determined by the investigator in consultation with the Amgen physician;

Exclusion Criteria:

- History or evidence of clinically significant disorder (including psychiatric), condition or disease that, in the opinion of the Investigator or Amgen physician would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2014-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Leuven, Belgium

REFERENCES:
- [Background] de Hoon J, Van Hecken A, Vandermeulen C, Yan L, Smith B, Chen JS, Bautista E, Hamilton L, Waksman J, Vu T, Vargas G. Phase I, Randomized, Double-blind, Placebo-controlled, Single-dose, and Multiple-dose Studies of Erenumab in Healthy Subjects and Patients With Migraine. Clin Pharmacol Ther. 2018 May;103(5):815-825. doi: 10.1002/cpt.799. Epub 2017 Oct 24. PMID 28736918
- [Derived] Kudrow D, Pascual J, Winner PK, Dodick DW, Tepper SJ, Reuter U, Hong F, Klatt J, Zhang F, Cheng S, Picard H, Eisele O, Wang J, Latham JN, Mikol DD. Vascular safety of erenumab for migraine prevention. Neurology. 2020 Feb 4;94(5):e497-e510. doi: 10.1212/WNL.0000000000008743. Epub 2019 Dec 18. PMID 31852816
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled healthy participants (Part A) and participants with onset of migraines before the age of 50 years, with or without aura for at least 6 months and 3 migraine attacks per month in the last 3 months (Part B). The study was conducted at a single center in Belgium.
Pre-assignment Details: Healthy participants were randomized to 1 of 4 cohorts and migraine patients were randomized to 1 of 2 cohorts. Within each cohort participants were assigned to erenumab or placebo in a 3:1 ratio.
Groups:
- Healthy: Placebo: Healthy participants received placebo subcutaneous injection on Days 1, 29, and 57.
- Healthy: Erenumab 21 mg: Healthy participants received 21 mg erenumab by subcutaneous injection on days 1, 29 and 57.
- Healthy: Erenumab 70 mg: Healthy participants received 70 mg erenumab by subcutaneous injection on days 1, 29 and 57.
- Healthy: Erenumab 140 mg: Healthy participants received 140 mg erenumab by subcutaneous injection on days 1, 29 and 57.
- Healthy: Erenumab 280/210 mg: Healthy participants received 280 mg erenumab by subcutaneous injection on day 1, and 210 mg erenumab on days 29 and 57.
- Migraine: Placebo: Participants with migraine received placebo by subcutaneous injection on days 1, 29 and 57.
- Migraine: Erenumab 21 mg: Participants with migraine received 21 mg erenumab by subcutaneous injection on days 1, 29 and 57.
- Migraine: Erenumab 140 mg: Participants with migraine received 140 mg erenumab by subcutaneous injection on days 1, 29 and 57.
Period: Overall Study
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Started | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are reported separately for each part of the study.
  years
    Healthy Participants: number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 32
    Healthy Participants | 32.1 (13.0) | 26.3 (5.7) | 33.3 (14.1) | 29.8 (8.6) | 39.0 (13.8) |  |  |  | 32.1 (11.6)
    Migraine Participants: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 6 | 16
    Migraine Participants |  |  |  |  |  | 37.0 (11.9) | 31.7 (11.0) | 31.3 (12.6) | 32.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 2 | 3 | 4 | 5 | 15
  Male | 8 | 6 | 5 | 6 | 4 | 1 | 2 | 1 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a causal relationship with study treatment. The definition of adverse events includes worsening of a pre-existing medical condition. Laboratory value changes that require treatment or adjustment in current therapy are considered adverse events.
  Teatment-related adverse events (TRAEs) are those assessed by the investigator as being possibly related to study drug.
  A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal
  * life-threatening (places the subject at immediate risk of death)
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
Time Frame: From first dose of study drug until a maximum of 168 days after last dose (225 days)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants
  Any adverse event | 5 | 6 | 6 | 6 | 4 | 4 | 6 | 6
  Serious adverse event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  AE leading to discontinuation of study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  AE leading to discontinuation from study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 1
  Treatment-related serious adverse events | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  TRAE leading to discontinuation of study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  TRAE leading to discontinuation from study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Suicidal Ideation and Behavior as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a measure of suicidal ideation and behavior. Ideation includes a wish to be dead or nonspecific thoughts about wanting to end life. Suicidal behavior includes actual attempts, interrupted or aborted attempts, and any preparatory acts.
Time Frame: From first dose of study drug until a maximum of 168 days after last dose (225 days)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants
  Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Developed Anti-erenumab Antibodies
Description: Participants who had a negative or no result at baseline and were antibody positive postbaseline.
  Blood samples were first tested for anti-erenumab binding antibodies, samples testing positive for binding antibodies were also tested for neutralizing antibodies.
Time Frame: From first dose of study drug until a maximum of 168 days after last dose (225 days)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants
  Binding antibodies | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0
  Neutralizing antibodies | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Erenumab
Description: Serum concentration of erenumab was analyzed using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1 (assessed from predose to day 28) and day 57 (assessed from predose up to day 225)
Population: All participants for whom at least 1 pharmacokinetic parameter or endpoint was adequately estimated and with available data at each time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 0 | 6 | 6
μg/mL
  Day 1 |  | 2.15 (0.914) | 6.26 (2.55) | 13.8 (4.00) | 24.9 (4.90) |  | 1.76 (0.741) | 11.0 (3.85)
  Day 57: number analyzed (Participants) | 0 | 6 | 5 | 6 | 6 | 0 | 6 | 6
  Day 57 |  | 2.60 (0.952) | 9.63 (3.60) | 23.7 (7.89) | 36.3 (6.18) |  | 2.00 (0.552) | 18.4 (5.98)

5. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Erenumab
Description: Serum concentration of erenumab was analyzed using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1 (assessed from predose to day 28) and day 57 (assessed from predose up to day 225)
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 0 | 6 | 6
days
  Day 1 |  | 4.0 [3.0 to 6.9] | 4.0 [3.0 to 11] | 5.9 [3.1 to 13] | 6.9 [3.0 to 6.9] |  | 6.9 [4.0 to 7.0] | 11 [4.0 to 13]
  Day 57: number analyzed (Participants) | 0 | 6 | 5 | 6 | 6 | 0 | 6 | 6
  Day 57 |  | 6.9 [5.9 to 7.9] | 7.9 [6.9 to 14] | 6.9 [6.9 to 8.0] | 6.9 [6.9 to 8.0] |  | 6.9 [6.9 to 7.9] | 6.9 [6.9 to 7.0]

6. Secondary Outcome: Area Under the Serum Concentration-Time Curve From 0 to 28 Days (AUC0-28day)
Description: Serum concentration of erenumab was analyzed using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1 (assessed from predose to day 28) and day 57 (assessed from predose up to day 225)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 0 | 6 | 6
day*μg/mL
  Day 1 |  | 34.7 (13.1) | 124 (49.2) | 281 (89.1) | 486 (57.8) |  | 28.7 (11.0) | 244 (86.2)
  Day 57: number analyzed (Participants) | 0 | 6 | 5 | 6 | 6 | 0 | 6 | 6
  Day 57 |  | 49.5 (20.1) | 216 (82.7) | 476 (161) | 760 (143) |  | 37.9 (12.5) | 417 (117)

7. Secondary Outcome: Area Under the Serum Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast)
Description: Serum concentration of erenumab was analyzed using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 57 (assessed from predose to day 225))
Population: All participants who received erenumab and for whom at least 1 pharmacokinetic parameter or endpoint was adequately estimated and with available data at each time point.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 0 | 6 | 6
day*μg/mL |  | 59.3 (27.8) | 342 (144) | 848 (376) | 1410 (332) |  | 45.0 (15.7) | 773 (214)

8. Secondary Outcome: Ratio of Post-capsaicin Dermal Blood Flow to Pre-capsaicin Dermal Blood Flow
Description: Inhibition of capsaicin-induced dermal blood flow (DBF) by erenumab was used to measure calcitonin gene-related peptide (CGRP) receptor antagonism. Capsaicin was applied at 2 sites on the volar surface of the participants' left or right forearms and a control mixture was applied to 1 site on the volar surface of either the participants' left or right forearm. Dermal blood flow was assessed by laser Doppler perfusion imaging and was done immediately before ('baseline') and 0.5 hours post-capsaicin on the surface of these 3 sites.
  Data reported are the least square geometric mean ratios for the post-capsaicin dermal blood flow to pre-capsaicin dermal blood flow.
  According to the protocol, not all cohorts had dermal blood flow measurements at all time points.
Time Frame: Baseline, Days 8, 57, 85, 113, 169 and 197
Population: All participants for whom at least 1 postdose capsaicin response measure was recorded. Measurement and analysis of dermal blood flow were not performed in the 280/210 cohort.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0 | 4 | 6 | 6
ratio
  Baseline | 9.24 (1.20) | 9.28 (1.21) | 8.92 (1.20) | 8.90 (1.22) |  | 13.27 (1.37) | 11.08 (1.29) | 11.70 (1.28)
  Day 8 | 8.53 (1.20) | 1.76 (1.21) | 2.46 (1.20) | 1.75 (1.22) |  | 13.20 (1.37) | 2.64 (1.29) | 1.64 (1.28)
  Day 57 | 6.75 (1.20) | 1.87 (1.21) | 1.82 (1.20) | 1.90 (1.22) |  | 12.30 (1.37) | 2.48 (1.29) | 2.01 (1.28)
  Day 85 | 8.61 (1.20) | 2.71 (1.21) | 1.63 (1.20) | 1.80 (1.22) |  | 13.33 (1.37) | 2.40 (1.29) | 2.08 (1.28)
  Day 113: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0 | 4 | 6 | 0
  Day 113 | 11.11 (1.33) | 7.48 (1.21) |  |  |  | 3.50 (1.51) | 5.00 (1.29) |
  Day 169: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 4 | 0 | 6
  Day 169 | 9.72 (1.24) |  | 10.06 (1.20) | 5.78 (1.22) |  | 14.78 (1.51) |  | 4.64 (1.28)
  Day 197: number analyzed (Participants) | 6 | 0 | 0 | 6 | 0 | 4 | 0 | 6
  Day 197 | 7.20 (1.33) |  |  | 8.16 (1.22) |  | 18.52 (1.51) |  | 8.46 (1.28)
Statistical Analysis 1: Comparison: Healthy: Placebo vs Healthy: Erenumab 21 mg; Day 8: A repeated measures ANCOVA was performed for the ratio of blood flow measures at 30 minutes post capsaicin challenge to pre capsaicin challenge. The model included treatment, day, and the treatment by day interaction as independent variables, and both the 0 minute pre-capsaicin blood flow measure as well as the day 0, 30-minute post-capsaicin blood flow measures on day -1; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -79.33, 95% CI 2-sided [-87.54 to -65.73]
Statistical Analysis 2: Comparison: Healthy: Placebo vs Healthy: Erenumab 70 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -71.16, 95% CI 2-sided [-82.67 to -52.00]
Statistical Analysis 3: Comparison: Healthy: Placebo vs Healthy: Erenumab 140 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -79.52, 95% CI 2-sided [-88.29 to -64.17]
Statistical Analysis 4: Comparison: Healthy: Placebo vs Healthy: Erenumab 21 mg; Day 57: A repeated measures ANCOVA was performed for the ratio of blood flow measures at 30 minutes post capsaicin challenge to pre capsaicin challenge. The model included treatment, day, and the treatment by day interaction as independent variables, and both the 0 minute pre-capsaicin blood flow measure as well as the day 0, 30-minute post-capsaicin blood flow measures on day -1; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -72.34, 95% CI 2-sided [-83.32 to -54.13]
Statistical Analysis 5: Comparison: Healthy: Placebo vs Healthy: Erenumab 70 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -73.03, 95% CI 2-sided [-83.79 to -55.11]
Statistical Analysis 6: Comparison: Healthy: Placebo vs Healthy: Erenumab 140 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -71.88, 95% CI 2-sided [-83.93 to -50.82]
Statistical Analysis 7: Comparison: Healthy: Placebo vs Healthy: Erenumab 21 mg; Day 85: A repeated measures ANCOVA was performed for the ratio of blood flow measures at 30 minutes post capsaicin challenge to pre capsaicin challenge. The model included treatment, day, and the treatment by day interaction as independent variables, and both the 0 minute pre-capsaicin blood flow measure as well as the day 0, 30-minute post-capsaicin blood flow measures on day -1; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -68.51, 95% CI 2-sided [-81.01 to -47.78]
Statistical Analysis 8: Comparison: Healthy: Placebo vs Healthy: Erenumab 70 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -81.06, 95% CI 2-sided [-88.62 to -68.49]
Statistical Analysis 9: Comparison: Healthy: Placebo vs Healthy: Erenumab 140 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -79.04, 95% CI 2-sided [-88.02 to -63.34]
Statistical Analysis 10: Comparison: Healthy: Placebo vs Healthy: Erenumab 21 mg; Day 113: A repeated measures ANCOVA was performed for the ratio of blood flow measures at 30 minutes post capsaicin challenge to pre capsaicin challenge. The model included treatment, day, and the treatment by day interaction as independent variables, and both the 0 minute pre-capsaicin blood flow measure as well as the day 0, 30-minute post-capsaicin blood flow measures on day -1; Test type: Superiority; p = 0.25, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -32.70, 95% CI 2-sided [-65.71 to 32.10]
Statistical Analysis 11: Comparison: Healthy: Placebo vs Healthy: Erenumab 70 mg; Day 169: A repeated measures ANCOVA was performed for the ratio of blood flow measures at 30 minutes post capsaicin challenge to pre capsaicin challenge. The model included treatment, day, and the treatment by day interaction as independent variables, and both the 0 minute pre-capsaicin blood flow measure as well as the day 0, 30-minute post-capsaicin blood flow measures on day -1; Test type: Superiority; p = 0.90, Repeated Measures ANCOVA; LS Geometric Mean Ratio = 3.44, 95% CI 2-sided [-40.78 to 80.66]
Statistical Analysis 12: Comparison: Healthy: Placebo vs Healthy: Erenumab 140 mg; [analysis description as in outcome 8, analysis 11]; Test type: Superiority; p = 0.091, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -40.53, 95% CI 2-sided [-67.50 to 8.82]
Statistical Analysis 13: Comparison: Healthy: Placebo vs Healthy: Erenumab 140 mg; Day 197: A repeated measures ANCOVA was performed for the ratio of blood flow measures at 30 minutes post capsaicin challenge to pre capsaicin challenge. The model included treatment, day, and the treatment by day interaction as independent variables, and both the 0 minute pre-capsaicin blood flow measure as well as the day 0, 30-minute post-capsaicin blood flow measures on day -1; Test type: Superiority; p = 0.73, Repeated Measures ANCOVA; LS Geometric Mean Ratio = 13.33, 95% CI 2-sided [-44.39 to 130.94]
Statistical Analysis 14: Comparison: Migraine: Placebo vs Migraine: Erenumab 21 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -80.02, 95% CI 2-sided [-91.53 to -52.87]
Statistical Analysis 15: Comparison: Migraine: Placebo vs Migraine: Erenumab 140 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -87.60, 95% CI 2-sided [-94.53 to -71.88]
Statistical Analysis 16: Comparison: Migraine: Placebo vs Migraine: Erenumab 21 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p = 0.001, Repeated Measures ANCOVA; LS Geometric Mean Rratio = -79.81, 95% CI 2-sided [-91.44 to -52.37]
Statistical Analysis 17: Comparison: Migraine: Placebo vs Migraine: Erenumab 140 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -83.66, 95% CI 2-sided [-92.79 to -62.95]
Statistical Analysis 18: Comparison: Migraine: Placebo vs Migraine: Erenumab 21 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -81.97, 95% CI 2-sided [-92.35 to -57.46]
Statistical Analysis 19: Comparison: Migraine: Placebo vs Migraine: Erenumab 140 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -84.39, 95% CI 2-sided [-93.12 to -64.60]
Statistical Analysis 20: Comparison: Migraine: Placebo vs Migraine: Erenumab 21 mg; [analysis description as in outcome 8, analysis 10]; Test type: Superiority; p = 0.47, Repeated Measures ANCOVA; LS Geometric Mean Ratio = 43.10, 95% CI 2-sided [-47.06 to 286.83]
Statistical Analysis 21: Comparison: Migraine: Placebo vs Migraine: Erenumab 140 mg; [analysis description as in outcome 8, analysis 11]; Test type: Superiority; p = 0.020, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -68.58, 95% CI 2-sided [-88.02 to -17.63]
Statistical Analysis 22: Comparison: Migraine: Placebo vs Migraine: Erenumab 140 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority; p = 0.11, Repeated Measures ANCOVA; LS Geometric Mean Ratio = -54.32, 95% CI 2-sided [-82.58 to 19.75]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until a maximum of 168 days after last dose (225 days).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Healthy: Placebo | Healthy: Erenumab 21 mg | Healthy: Erenumab 70 mg | Healthy: Erenumab 140 mg | Healthy: Erenumab 280/210 mg | Migraine: Placebo | Migraine: Erenumab 21 mg | Migraine: Erenumab 140 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 1/6 | 0/6 | 0/6 | 0/4 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 5/8 | 6/6 | 6/6 | 6/6 | 4/6 | 4/4 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy: Placebo (N=8) | Healthy: Erenumab 21 mg (N=6) | Healthy: Erenumab 70 mg (N=6) | Healthy: Erenumab 140 mg (N=6) | Healthy: Erenumab 280/210 mg (N=6) | Migraine: Placebo (N=4) | Migraine: Erenumab 21 mg (N=6) | Migraine: Erenumab 140 mg (N=6)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy: Placebo (N=8) | Healthy: Erenumab 21 mg (N=6) | Healthy: Erenumab 70 mg (N=6) | Healthy: Erenumab 140 mg (N=6) | Healthy: Erenumab 280/210 mg (N=6) | Migraine: Placebo (N=4) | Migraine: Erenumab 21 mg (N=6) | Migraine: Erenumab 140 mg (N=6)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Influenza like illness (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 3 | 0 | 1 | 1 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2 | 3 | 0 | 0 | 3 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 3 | 2 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood immunoglobulin E increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 3 | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.